CLINICAL TRIAL: NCT01132586
Title: Phase I Study of Lenalidomide and Conventional Chemotherapy in Acute Myeloid Leukemia
Brief Title: Lenalidomide, Cytarabine, and Idarubicin in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01375; NCI-2011-01375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA076576 (NIH); OSU-10016; CDR0000673883; OSU 10016 (Other: Ohio State University Comprehensive Cancer Center); 8455 (Other: CTEP); UM1CA186712 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-11

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Promyelocytic Leukemia With t(15;17)(q22;q12); PML-RARA; Alkylating Agent-Related Acute Myeloid Leukemia; de Novo Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndrome; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Acute | interventions — Lenalidomide; Cytarabine; Idarubicin; 4-demethoxydaunorubicin bis(hydrazone)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide, cytarabine, idarubicin) (Experimental): INDUCTION:
  COHORT I: Patients receive lenalidomide PO QD on days 1-21, cytarabine IV continuously over 96 hours on days 5-8, and idarubicin IV over 1 hour on days 5-7.
  COHORT II: Patients receive lenalidomide PO QD on days 1-21, cytarabine IV continuously over 24 hours on days 5-11, and idarubicin as above.
  Patients with residual disease on day 18 undergo a second course of induction therapy.
  CONSOLIDATION:
  COHORT I: Patients receive lenalidomide PO QD on days 1-14, idarubicin IV over 1 hour on days 5-6, cytarabine IV continuously on days 5-7. Treatment continues for 1 course in the absence of disease progression or unacceptable toxicity.
  COHORT II: Patients 2 receive 4 courses of consolidation therapy comprising lenalidomide PO QD on days 1-14 and cytarabine IV every 12 hours on days 5, 7, and 9. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Drug: Cytarabine; Drug: Idarubicin; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; IMiD-1
Drug: Cytarabine — Given IV
  Other Names: CHX-3311; U-19920
Drug: Idarubicin — Given IV
  Other Names: Idamycin; IMI-30; SC-33428; Zavedos
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with cytarabine and idarubicin in treating patients with acute myeloid leukemia. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as cytarabine and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with cytarabine and idarubicin may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of lenalidomide in combination with conventional chemotherapy in two separate cohorts of patients with 1) relapsed or refractory acute myeloid leukemia (AML) and 2) age >= 60 with untreated AML and recommend starting doses for phase II studies of this combination of agents.

SECONDARY OBJECTIVES:

I. To define the qualitative and quantitative toxicities of these combinations of agents in regard to organ specificity, time course, predictability, and reversibility.

II. To document the therapeutic response of these combinations of agents in patients with poor risk AML.

III. To conduct pharmacodynamic studies to investigate the potential mechanism of lenalidomide activity in this trial.

OUTLINE: This is a dose-escalation study of lenalidomide.

INDUCTION:

COHORT I: Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21, cytarabine intravenously (IV) continuously over 96 hours on days 5-8, and idarubicin IV over 1 hour on days 5-7.

COHORT II: Patients receive lenalidomide PO QD on days 1-21, cytarabine IV continuously over 24 hours on days 5-11, and idarubicin as above.

Patients with residual disease on day 18 undergo a second course of induction therapy.

CONSOLIDATION:

COHORT I: Patients receive lenalidomide PO QD on days 1-14, idarubicin IV over 1 hour on days 5-6, cytarabine IV continuously on days 5-7. Treatment continues for 1 course in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients 2 receive 4 courses of consolidation therapy comprising lenalidomide PO QD on days 1-14 and cytarabine IV every 12 hours on days 5, 7, and 9. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Patients must be age >= 18 and < 65 with relapsed or refractory AML or high risk myelodysplastic syndrome (MDS); high risk MDS is defined as international prognosis scoring system (IPSS) score of 1.5 or higher; eligible patients will have a score of 1.5 or higher at any time from diagnosis to screening

  * Cohort 2: Patients must be age >= 18 with previously untreated AML; favorable risk AML patients < 60 years of age are excluded; these are defined as core binding factor (CBF) AML patients and characterized by cytogenetic or molecular evidence of CBF leukemia; untreated AML patients < 60 years of age must be negative on screening for CBF leukemia by cytogenetic or molecular analysis (Note: Prior therapy for MDS is permitted)
* Patients with secondary AML or therapy-related disease (transformed [t]-AML/MDS) are eligible
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2.5 times upper limit of normal
* Creatinine < 2.0 mg/dL AND creatinine clearance (calculated) >= 50 mL/min
* Left ventricular ejection fraction (LVEF) >= 40%
* Patients who have previously received lenalidomide, idarubicin, and/or cytarabine are eligible provided that the combination of the 3 agents has never before been administered, and that no lenalidomide has been administered for at least 6 months
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a minimum sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; these methods of birth control must be used for the duration of study participation and for 28 days after lenalidomide discontinuation; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Ability to understand and willingness to sign the written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have taken lenalidomide within the last 6 months
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system disease or with granulocytic sarcoma as sole site of disease
* Patients with history of medically serious allergic reactions or non-hematologic toxicities attributed to the agents in this trial such as lenalidomide or thalidomide or compounds of similar chemical or biologic composition that are not easily managed, or patients with a history of cerebellar toxicity to cytarabine
* Patients with the following will be excluded: uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; patients with medical comorbidities that will preclude safety evaluation of the combination should not be enrolled
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding; additional pregnancy testing before, during, and after lenalidomide treatment is required, as well as requirements for contraception before, during, and after lenalidomide treatment
* Patients with advanced malignant solid tumors are excluded; patients with active additional hematologic malignancies are excluded
* Patients with a history of neurologic toxicity with cytarabine are excluded
* As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control; patients with uncontrolled infection shall not be enrolled until infection is treated and brought under control
* Known human immunodeficiency virus (HIV)-positive patients are ineligible; appropriate studies will be undertaken in HIV + patients once safety of the combination has been demonstrated

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide, determined according to incidence of dose-limiting toxicity (DLT) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 28 days

SECONDARY OUTCOMES:
Qualitative and quantitative toxicities, graded using NCI CTCAE version 4.0 | Up to 30 days post-treatment
Therapeutic response, assessed using International Working Group criteria | Up to 30 days post-treatment
Pharmacodynamic studies, including micro-ribonucleic acid (miRNA)-181 family and target gene expression, CCAAT/enhancer binding protein (C/EBP), alpha gene (CEBPA) expression, and genes involved in erythroid differentiation | Baseline, day 5, and day 28

CONTACTS AND LOCATIONS:
Overall Officials: William Blum, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Saygin C, Larkin K, Blachly JS, Orwick S, Ngankeu A, Gregory CT, Phelps MA, Mani S, Walker A, Garzon R, Vasu S, Walsh KJ, Bhatnagar B, Klisovic RB, Grever MR, Marcucci G, Byrd JC, Blum W, Mims AS. A phase I study of lenalidomide plus chemotherapy with idarubicin and cytarabine in patients with relapsed or refractory acute myeloid leukemia and high-risk myelodysplastic syndrome. Am J Hematol. 2020 Dec;95(12):1457-1465. doi: 10.1002/ajh.25958. Epub 2020 Sep 19. PMID 32777116